CLINICAL TRIAL: NCT05774067
Title: Noradrenaline Versus Glypressin for Prevention of Hypotension After Deflation of Tourniquet in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: tourniquet deflation
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Norepinephrine, Glypressin, Tourniquet Deflation; Hypotension
MeSH Terms: conditions — Hypotension | interventions — Sodium Chloride; Norepinephrine; Terlipressin; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator)
  Interventions: Drug: Saline
- noradrenaline (Active Comparator)
  Interventions: Drug: Norepinephrine
- glypressin (Active Comparator)
  Interventions: Drug: glypressin

INTERVENTIONS:
Drug: Saline — patient received normal saline 4ml/kg/hr with deflation of tourniquet
  Other Names: control
  Arms: control
Drug: Norepinephrine — patient received noradrenaline infusion at rate 0.1 mcg/kg/min. with deflation of tourniquet
  Other Names: noradrenaline
  Arms: noradrenaline
Drug: glypressin — patient receive glypressin infusion at rate 2 mcg/kg/hr.
  Other Names: vasopressin
  Arms: glypressin

SUMMARY:
Pneumatic tourniquet is usually used in orthopedic surgeries, as it helps to decrease operative bed bleeding, and thus, maintaining a clean and dry surgical field allowing easy and clear identification of the anatomical structures. Despite that advantage, after its deflation, there is a blood volume shift towards that ischemic area, which may decrease cardiac preload leading to hypotension

DETAILED DESCRIPTION:
Hemodynamic changes after tourniquet deflation include; hypotension, tachycardia and increase in cardiac index. These changes may be insignificant for healthy individuals but, risky for patients with compromised cardiovascular system and geriatric population.

Hypovolemia is a common problem in many clinical situations. The mortality of hypovolemic shock is directly related to the severity and duration of organ hypoperfusion.

Management of hypotension include frequent monitoring of blood pressure, fluid therapy, non-pharmacological methods, and vasopressors. Fluid therapy by crystalloids or colloids has been the traditional approach to restore volume and can be given as preload or co-load .Non pharmacological methods include positioning and leg compression. Trendelenburg position can increase venous return to the heart. Leg compression by flexion of the hip, elastic bandages, or stockings. An efficient method to treat spinal hypotension is administration of vasopressors, either given by infusion or boluses. Vasopressor drugs act by reversing the circulatory effect of sympathetic blockade. They also restore vascular tone and preserve venous return and cardiac filling

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients of both gender
* American Society of Anesthesiologists (ASA) I or II
* scheduled for elective unilateral total knee arthroplasty

Exclusion Criteria

* Patient refusal.
* Major cardiopulmonary disorders
* Uncontrolled systemic hypertension.
* Hepatic or renal disorders.
* Patient with relative contraindication for tourniquet use as peripheral vascular disease, sickle cell anemia, deep venous thrombosis, diabetic neuropathy and crushed injury.
* Cases having American Society of Anesthesiologists [ASA] > II
* Coagulopathy and bleeding tendency.
* Revision knee arthroplasty and bilateral knee arthroplasty

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
change of mean arterial blood pressure | 30 minutes after tourniquet deflation
  change of mean arterial bllod pressure till 30 min after deflation of the tourniquet.

CONTACTS AND LOCATIONS:
Overall Officials: reda sobhy, MD, Study Director — tanta university, faculty of medicine
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No